CLINICAL TRIAL: NCT01931150
Title: A Phase III Randomized Double-blind Study of Prophylactic Topical Dapsone 5% Gel Versus Moisturizer for Cetuximab-induced Papulopustular (Acneiform) Rash in Patients With mCRC or HNSCC Without Previous or Concurrent RT
Brief Title: Study of Prophylactic Topical Dapsone 5% Gel Versus Moisturizer for Cetuximab-induced Papulopustular (Acneiform) Rash in Patients With mCRC or HNSCC Without Previous or Concurrent RT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-012
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Cetuximab-induced Papulopustular (Acneiform) Rash Who Have; Metastatic Colorectal Cancer or Head and Neck Squamous Cell Carcinoma
Keywords: Topical Dapsone 5% Gel; Moisturizer; rash; 13-012
MeSH Terms: conditions — Colorectal Neoplasms; Exanthema | interventions — Dapsone; Gels; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dapsone LEFT, Moisturizer RIGHT (Experimental): Dapsone 5% gel to LEFT side of face and chest BID (morning and evening) Moisturizer to RIGHT side of face and chest BID (morning and evening) AND oral antibiotics (doxycycline 100 mg bid OR minocycline 100 mg once daily or other antibiotic daily)
  Interventions: Drug: Topical Dapsone 5% Gel; Other: Moisturizer; Drug: oral antibiotics
- Dapsone RIGHT, Moisturizer LEFT (Experimental): Moisturizer to LEFT side of face and chest BID (morning and evening) Dapsone 5% gel to RIGHT side of face and chest BID (morning and evening) AND oral antibiotics (doxycycline 100 mg bid OR minocycline 100 mg once daily or other antibiotic daily)
  Interventions: Drug: Topical Dapsone 5% Gel; Other: Moisturizer; Drug: oral antibiotics

INTERVENTIONS:
Drug: Topical Dapsone 5% Gel
Other: Moisturizer — The moisturizer for the study will be Vanicream™ Lite Lotion.
Drug: oral antibiotics

SUMMARY:
The purpose of this study is to see if the investigators can prevent or reduce the severity of the Cetuximab-related acne rash. Two different topical agents will be applied to the skin. One topical agent is the dapsone gel and the other is a skin moisturizer. Dapsone gel is an FDA approved medication that you apply to the face. It is commonly used to treat acne. Skin moisturizers are recommended to patients who receive Cetuximab treatment. In addition to these topical agents they will be given a pill to take once a day. This pill has already been shown to help fight rashes from Cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with underlying diagnosis of metastatic colorectal cancer or head and neck squamous cell carcinoma including newly diagnosed patient
* Patients must provide written informed consent to participate in the study
* Anticipated initiation of cetuximab treatment with or without additional chemotherapy.
* Able to self-administer topical interventions or provide for another person to apply the topical interventions

Exclusion Criteria:

* Females of childbearing potential who are pregnant or nursing
* Patients with allergy, hypersensitivity or other contraindication to dapsone, sulfa antibiotics, or excipients of the dapsone gel product
* Patients with pre-existing dermatologic condition affecting the face and chest that would impair assessment of papulopustular rash including dense and/or long facial hair (per investigator discretion)
* Patients currently using prescription and/or over-the-counter topical medications to the face and/or chest who are unwilling to discontinue use during the trial intervention period (day 0 ± 2 days through day 28 ± 2 days)
* Previous or concurrent radiation therapy to head, neck, and chest (i.e. application sites only)
* Previous therapy with cetuximab within 6 months of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Lacouture, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapsone LEFT, Moisturizer RIGHT: Arm1: Receive oral antibiotics AND apply Dapsone 5% gel to LEFT side of face and chest BID (morning and evening), AND moisturizer to RIGHT side of face and chest BID (morning and evening), for 28 +/- 2 days.
- Dapsone RIGHT, Moisturizer LEFT: Arm 2: Receive oral antibiotics AND apply Dapsone 5% to RIGHT side of face and chest BID (morning and evening), AND moisturizer to LEFT side of face and chest BID (morning and evening), for 28 +/- 2 days.
Period: Overall Study
Arm/Group | Dapsone LEFT, Moisturizer RIGHT | Dapsone RIGHT, Moisturizer LEFT
Started | 5 | 6
Completed | 4 | 4
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapsone LEFT, Moisturizer RIGHT | Dapsone RIGHT, Moisturizer LEFT | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 1 | 1
Gender [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Which the PI Observed a Notable Difference in the Number of Lesions
Description: Change from Baseline in the Number of Lesions at 28 days
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Dapsone LEFT, Moisturizer RIGHT | Dapsone RIGHT, Moisturizer LEFT
Number analyzed (Participants) | 4 | 4
participants | 4 | 4

ADVERSE EVENTS:
Arm/Group | Dapsone LEFT, Moisturizer RIGHT | Dapsone RIGHT, Moisturizer LEFT
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapsone LEFT, Moisturizer RIGHT (N=5) | Dapsone RIGHT, Moisturizer LEFT (N=6)
Allergic reaction (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes